CLINICAL TRIAL: NCT02047396
Title: Ventricular Remodeling and Heart Failure After Myocardial Infarction: a Community Study
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Suzette J. Bielinski, Principal Investigator, Mayo Clinic
Other Study IDs: 13-009187; R01HL136659 (NIH)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Myocardial Infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, and WBCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial Infarction subjects: Subjects with first Myocardial Infarction presenting to one of the Mayo Clinic Hospitals in Rochester, Minnesota.

SUMMARY:
To comprehensively characterize Left Ventricular (LV) remodeling after Myocardial Infarction (MI) in the community, study the association between patterns of remodeling and biological pathways and examine the association between the predictors of remodeling and heart failure after Myocardial Infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with a clinical diagnosis of Myocardial Infarction.
2. Residents of Olmsted, Dodge, Goodhue, Wabasha, Winona, Fillmore and Mower Counties.
3. Able to provide informed consent.

Exclusion Criteria:

1. Previous clinical diagnosis of Myocardial Infarction
2. Previous diagnosis of Heart Failure and/or Cardiomyopathy
3. Diagnosis of Apical Ballooning Syndrome
4. Planned Coronary Artery Bypass Graft (CABG) during index hospitalization
5. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in the 7 County area who are admitted to the Mayo Clinic Hospitals in Rochester, Minnesota who have their first myocardial infarction and are willing to have blood drawn and return for an echocardiogram in 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 1599 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Heart Failure | 5 years
  Development of Heart Failure post Myocardial Infarction

SECONDARY OUTCOMES:
Death | 5 years
  All cause mortality post Myocardial Infarction

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Bielinski, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No